CLINICAL TRIAL: NCT04104061
Title: Iron Profile in Patients With Congenital Cyanotic Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Sami Abdelrahman, principal investigator, Assiut University
Other Study IDs: ipipwcchd
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Congenital; Cyanotic Heart Disease
MeSH Terms: interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: iron profile — blood test
  Other Names: complete blood count

SUMMARY:
Iron is a vital substrate for hemoglobin production and sufficient iron stores are necessary to achieve and maintain adequate levels of hemoglobin.

DETAILED DESCRIPTION:
Iron is a vital substrate for hemoglobin production and sufficient iron stores are necessary to achieve and maintain adequate levels of hemoglobin. Unfortunately, more than one third of patients with cyanotic heart disease are iron-deficient (1),(2). In 1990, West et al, have demonstrated that more than one-third of patients with congenital cyanotic heart diseases (CCHD) had iron deficiency(3) In another study done by Olcay et al, the prevalence of iron deficiency anemia (IDA) was found to be 52.2%(4).

Possible causes of iron deficiency include increased iron consumption through increased erythropoiesis, inappropriate venesections, hemoptysis, bleeding from arteriovenous malformations or collateral vessels, abnormal hemostasis, limited dietary intake or absorption, and use of anticoagulants and antiplatelets (5).

Also congenital cyanotic heart lesions are associated with a state of constant hypoxia This hypoxia triggers a physiological increase in erythropoietin release leading to stimulation of the bone marrow to produce more red cells in an effort to increase the body's oxygen carrying capacity, so as to improve oxygen delivery to the tissues. With persisting right to left shunt, the arterial oxygen tensions remain perpetually low and so the production of more and more red cells goes unabated leading to polycythemia. This seemingly noble physiological response eventually leads to depletion of iron stores (6).

In these patients, the total haemoglobin is normal, high or slightly reduced compared to aged-matched normal individuals without cyanosis. However, the MCV, MCH and serum ferritin are usually comparatively lower than their peers as shown by Cemile et al - a phenomenon known as relative anemia (7).

In fact, traditional diagnostic criteria for anemia do not apply to these patients, where "appropriate" levels of hemoglobin may vary according to their oxygen saturations (8). Also, other erythrocyte indices such as MCV and MCH are not sensitive indicators of iron deficiency in cyanotic patients (9).

IDA aggravates hyperviscosity symptoms due to the presence of microcytic erythrocytes not amenable to deformation in the microcirculation. Thus, presence of IDA in these children further increases their chances of morbidity in the form of cerebrovascular events and cyanotic spells (10).

The high incidence of iron deficiency among children with CCHD draws attention to the importance of evaluating iron deficiency in this population.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age: 1month to 18 years 2. Pediatric patients attending and admitted to Assuit University Children Hospital and diagnosed to have congenital cyanotic heart disease evidenced by clinical picture and echocardiography.

3. Both sexes.

Exclusion Criteria:

* 1. Patients with acyanotic congenital heart disease. 2. Patients who had surgical correction. 3. Patients who received iron supplements in previous three months. 4. Patients who have another systemic disease that affect iron profile and cause anemia as Chronic kidney disease or Hemolytic anemia

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: infants and n with congenital cyanotic heart disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
iron profile in patients with congenital cyanotic heart disease | 1 year
  iron profile in patients with congenital cyanotic heart disease

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mukherjee S, Sharma M, Devgan A, Jatana SK. Iron deficiency anemia in children with cyanotic congenital heart disease and effect on cyanotic spells. Med J Armed Forces India. 2018 Jul;74(3):235-240. doi: 10.1016/j.mjafi.2017.07.003. Epub 2017 Aug 18. PMID 30093766
- [Background] Lang'o MO, Githanga JN, Yuko-Jowi CA. Prevalence of iron deficiency in children with cyanotic heart disease seen at Kenyatta National Hospital and Mater Hospital Nairobi. East Afr Med J. 2009 Dec;86(12 Suppl):S47-51. doi: 10.4314/eamj.v86i12.62901. PMID 21591509
- [Result] Tay EL, Peset A, Papaphylactou M, Inuzuka R, Alonso-Gonzalez R, Giannakoulas G, Tzifa A, Goletto S, Broberg C, Dimopoulos K, Gatzoulis MA. Replacement therapy for iron deficiency improves exercise capacity and quality of life in patients with cyanotic congenital heart disease and/or the Eisenmenger syndrome. Int J Cardiol. 2011 Sep 15;151(3):307-12. doi: 10.1016/j.ijcard.2010.05.066. Epub 2010 Jul 1. PMID 20580108